CLINICAL TRIAL: NCT06657105
Title: An Open-label, Fixed Sequence Study to Assess the Effect of Multiple Doses of Baxdrostat on the Pharmacokinetics of Single Doses of Combined Oral Ethinyl Estradiol and Levonorgestrel in Healthy Female Participants of Non-childbearing Potential.
Brief Title: A Study to Investigate the Pharmacokinetics of Ethinyl Estradiol and Levonorgestrel When Given Alone and in Combination With Baxdrostat in Healthy Females of Non-childbearing Potential
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: D6970C00006
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Healthy Participants
Keywords: Baxdrostat; Aldosterone; Ethinyl estradiol/ Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Period 1: Ethinyl estradiol/Levonorgestrel (EE/LNG) (Experimental): Participants will receive oral dose of EE/LNG in the fasted state on Day ,1 followed by PK sampling of EE/LNG for 120 hours (EE 72 hours and LNG 120 hours).
  Interventions: Drug: EE/LNG
- Period 2: Baxdrostat (Experimental): Participants will self-administer the baxdrostat tablet once a day from Day 6 to Day 16.
  Interventions: Drug: Baxdrostat
- Period 3: Baxdrostat + EE/LNG (Experimental): Participants will receive baxdrostat once daily on Day 17 to Day 22 and will receive EE+LNG in the fasted state on Day 18, followed by oral dose of EE/LNG PK sampling for 120 hours (EE=72 hours and LNG=120 hours).
  Interventions: Drug: EE/LNG; Drug: Baxdrostat

INTERVENTIONS:
Drug: EE/LNG — EE/LNG tablet will be administered orally.
  Arms: Period 1: Ethinyl estradiol/Levonorgestrel (EE/LNG); Period 3: Baxdrostat + EE/LNG
Drug: Baxdrostat — Baxdrostat tablet will be administered orally.
  Arms: Period 2: Baxdrostat; Period 3: Baxdrostat + EE/LNG

SUMMARY:
The main purpose of the study is to assess the effect of multiple doses of baxdrostat on the pharmacokinetics (PK) of a single dose of combined oral ethinyl estradiol (EE) and levonorgestrel (LNG). Safety and tolerability of baxdrostat will be assessed during the study.

DETAILED DESCRIPTION:
This is an open-label, 3-period fixed sequence study conducted at a single Clinical Unit.

The study will comprise of:

* A Screening period of maximum 28 days.
* Period 1: - From Day -1 to Day 5.
* Period 2: -From Day 6 to Day 16
* Period 3: - From Day 17 to Day 23.
* A Final Follow-up Visit, 7 (± 2) days after the last PK sample in Period 3.

ELIGIBILITY:
Inclusion Criteria:

* Females must have a negative pregnancy test at the Screening Visit and Study Day -1 (admission to Clinical Unit) and must not be lactating and must be of non-childbearing potential, confirmed at Screening by fulfilling one of the following criteria:

  1. Postmenopausal defined as amenorrhea for at least 12 months following cessation of all exogenous hormonal treatments and FSH levels in the postmenopausal range (Follicular Stimulating Hormone (FSH) > 40 mIU/mL).
  2. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy but not tubal ligation or tubal occlusion.
* Have a Body Mass Index (BMI) between 18 and 30 kg/m2

Exclusion Criteria:

* History of any clinically important disease or disorder which, in the opinion of the Investigator
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Sex hormone therapy within one month before study.
* History of drug-related hepatic toxicity.
* History or family history of potential risk of arterial and venous thromboembolic events (eg, factor V Leiden mutation).
* History of cardiovascular risk (eg, history of myocardial infarction).
* Any laboratory values with the following deviations at the Screening Visit and Study Day -1 (admission to Clinical Unit).
* Any positive result on screening for serum HBsAg, HBcAb, HCV or HIV.
* History of any treatment with QT prolongation drugs.
* Current smokers or know history of alcohol or drug abuse.
* History or ongoing severe allergy/hypersensitivity.
* An increased risk for developing SAEs or a contraindication associated with administration of EE, or LNG such as history of thrombosis or thromboembolism, presence of estrogen dependent tumors, hypertension, migraines, and liver disease.
* Participants treated with strong CYP3A4 inhibitors or inducers within 3 months or longer (5 half-lives) prior to first administration of IMP in this study.
* Plasma donation within one month of the Screening Visit or any blood donation/blood loss > 500 mL during the 3 months prior to the Screening Visit.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 30 days or 5 half-lives (whichever is longest) of the first administration of IMP in this study.
* Participants who are vegans or have medical dietary restrictions and vulnerable participants.

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 22 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Area under concentration-time curve from time zero to infinity (AUCinf) | EE: Up to Day 21, LNG: Up to Day 23
  To assess the effect of multiple doses of baxdrostat on the PK of a single dose of combined oral EE/LNG in healthy females of non-childbearing potential.
Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) | EE: Up to Day 21, LNG: Up to Day 23
  To assess the effect of multiple doses of baxdrostat on the PK of a single dose of combined oral EE/LNG in healthy females of non-childbearing potential.
Maximum observed drug concentration (Cmax) | EE: Up to Day 21, LNG: Up to Day 23
  To assess the effect of multiple doses of baxdrostat on the PK of a single dose of combined oral EE/LNG in healthy females of non-childbearing potential.

SECONDARY OUTCOMES:
Maximum observed drug concentration (Cmax) of EE/LNG | EE: Up to Day 21, LNG: Up to Day 23
  To describe the PK of a single dose of combined oral EE and LNG in healthy females of non-childbearing potential.
Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) of EE/LNG | EE: Up to Day 21, LNG: Up to Day 23
  To describe the PK of a single dose of combined oral EE and LNG in healthy females of non-childbearing potential.
Area under concentration-time curve from time zero to infinity (AUCinf) of EE/LNG | EE: Up to Day 21, LNG: Up to Day 23
  To describe the PK of a single dose of combined oral EE and LNG in healthy females of non-childbearing potential.
Time to reach maximum observed concentration (tmax) | EE: Up to Day 21, LNG: Up to Day 23
  To describe the PK of a single dose of combined oral EE and LNG in healthy females of non-childbearing potential.
Terminal elimination half-life (t1/2λz) | EE: Up to Day 21, LNG: Up to Day 23
  To describe the PK of a single dose of combined oral EE and LNG in healthy females of non-childbearing potential.
Terminal rate constant (λz) | EE: Up to Day 21, LNG: Up to Day 23
  To describe the PK of a single dose of combined oral EE and LNG in healthy females of non-childbearing potential.
Ratio of EE or LNG to EE (alone) or LNG (alone) based on AUCinf (RAUCinf) | EE: Up to Day 21, LNG: Up to Day 23
  To describe the PK of a single dose of combined oral EE and LNG in healthy females of non-childbearing potential.
Ratio of EE or LNG to EE (alone) or LNG (alone) based on AUClast (RAUClast) | EE: Up to Day 21; LNG: Up to Day 23
  To describe the PK of a single dose of combined oral EE and LNG in healthy females of non-childbearing potential.
Ratio of EE or LN to EE (alone) or LNG (alone) based on Cmax (RCmax) | EE: Up to Day 21; LNG: Up to Day 23
  To describe the PK of a single dose of combined oral EE and LNG in healthy females of non-childbearing potential.
Number of participants with adverse event (AEs) | From screening (Day -28 to Day -2) to 8.5 weeks
  To examine the safety and tolerability of baxdrostat alone and in combination with combined oral EE and LNG.
Maximum observed drug concentration (Cmax) of Baxdrostat | Baxdrostat: Day 18 to Day 22
  To assess the PK of baxdrostat in healthy female participants of non-childbearing potential.
Observed lowest concentration before the next dose is administered (Day 22 pre-dose) (Ctrough) | Baxdrostat: Day 18 to Day 22
  To assess the PK of baxdrostat in healthy female participants of non-childbearing potential.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Brooklyn, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-leveldata from AstraZeneca group of companies sponsored clinical trials via therequest portal Vivli.org. All requests will be evaluated as per the AZ disclosurecommitment:https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure."Yes",indicates that AZ are accepting requests for IPD, but this does not mean allrequests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/